CLINICAL TRIAL: NCT04429152
Title: ADORE: A Single-arm, Phase 3, Pilot Study Investigating the Efficacy of Doravirine in Adults Living With HIV Experiencing Virological Failure on First-line Efavirenz-based Antiretroviral Therapy With Non-nucleoside Reverse Transcriptase Inhibitor Resistance
Brief Title: ADORE: Efficacy of DORavirine in Adults Living With HIV Experiencing Virological Failure on First-line Efavirenz-based Antiretroviral Therapy With NNRTI Resistance
Acronym: ADORE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor Francois Venter (Other)
Responsible Party: Sponsor-Investigator, Professor Francois Venter, Divisional Director: Ezintsha, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZMiM018
Record Dates: First submitted 2020-06-05; First posted 2020-06-12 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: HIV-1-infection
Keywords: Virological failure, first-line antiretroviral therapy; Doravirine; Delstrigo
MeSH Terms: interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doravirine (Experimental): Once-daily, fixed-dose combination of doravirine 100 mg, lamivudine 300 mg, and tenofovir disoproxil fumarate 300 mg (DOR/3TC/TDF).
  Interventions: Drug: Doravirine/Lamivudine/Tenofovir

INTERVENTIONS:
Drug: Doravirine/Lamivudine/Tenofovir — DOR/3TC/TDF 100/300/300 mg once daily fixed-dose combination
  Other Names: Delstrigo

SUMMARY:
This is a pilot study investigating the efficacy of Doravirine (DOR) in combination with Lamivudine (3TC) and Tenofovir Disoproxil Fumarate (TDF) administered over 48 weeks in adults living with HIV-1 experiencing virological failure on first-line Efavirenz-based antiretroviral therapy with non-nucleoside reverse transcriptase inhibitor resistance

DETAILED DESCRIPTION:
This is a single-arm, phase 3 pilot study investigating the efficacy of Doravirine (DOR) in combination with Lamivudine (3TC) and Tenofovir Disoproxil Fumarate (TDF) administered over 48 weeks in adults living with HIV-1 experiencing virological failure on first-line Efavirenz-based antiretroviral therapy with non-nucleoside reverse transcriptase inhibitor resistance.

Approximately 25 male and female participants 18 years and older infected with HIV-1 and experiencing virological failure on efavirenz-based ART will be administered a once-daily, fixed-dose combination of doravirine 100 mg, lamivudine 300 mg, and tenofovir disoproxil fumarate 300 mg (DOR/3TC/TDF). The study includes screening and baseline visits, 4 study visits from Week 4 to Week 36, and an end of study visit at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Adults living with HIV-1, 18 years and older
* Viral load 5000 - 60 000 copies/mL on first-line efavirenz-based antiretroviral therapy
* HIV genotype resistance test with first generation NNRTI resistance (e.g. K103N, Y181C, etc as listed in the protocol)
* CD4 > 200 cells/uL
* Creatinine clearance > 50 mL/min
* Body mass ≥ 35 kg.

Exclusion Criteria:

* Resistance to TDF on genotype (K65R)
* "Significant resistance" to doravirine, denoted by a Stanford Score ≥ 15 on genotype
* Virologic failure on any other regimen
* Women who are pregnant at the time of the screening or enrolment visits
* Active tuberculosis and/or are on anti-tuberculous therapy at the time of the screening or enrolment visits
* Taking and cannot discontinue prohibited concomitant medications listed in protocol at least two weeks prior to the enrolment visit and for the duration of the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with undetectable plasma HIV-1 RNA levels (<50 copies/mL) at week 24 | 24 weeks
  The proportion of participants with undetectable plasma HIV-1 RNA levels at Week 24 will be recorded.

SECONDARY OUTCOMES:
Proportion of patients with undetectable plasma HIV-1 RNA levels (<50 copies/mL) at weeks 4, 12 and 48 | At week 4, 12, 48
  Evaluation of viral suppression by recording the proportion of patients with undetectable plasma HIV-1 RNA levels (<50 copies/mL) at weeks 4, 12 and 48
Change from baseline in plasma CD4 levels at weeks 24 and 48 | At week 24, 48
  Evaluation of changes in CD4 count from baseline recorded at weeks 24 and 48.
Emergence of antiretroviral resistance mutations in participants with virological failure | 48 weeks
  Evaluation of the number of antiretroviral resistance mutations that emerge in participants with virological failure

CONTACTS AND LOCATIONS:
Overall Officials: Simiso Sokhela, MBBCh, Principal Investigator — Ezintsha, a subdivision of Wits Reproductive Health and HIV Institute (Wits RHI)
Locations (3):
- South Africa (3):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Sunnyside Office Park, Johannesburg, Gauteng
  - Wits RHI Yeoville Clinic, Johannesburg, Gauteng